CLINICAL TRIAL: NCT01080625
Title: Effect of Preventive Medicine on the Postreperfusion Syndrome
Brief Title: Effect of Epinephrine/ Phenylephrine for Preventing the Postreperfusion Syndrome During Reperfusion in Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Assistant professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CWJung_phen_epi_liver TPL
Record Dates: First submitted 2010-03-02; First posted 2010-03-04 (Estimated); Results first posted 2012-04-12 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Hypotension After Reperfusion in Liver Transplantation
Keywords: postreperfusion syndrome; phenylephrine; epinephrine; liver transplantation
MeSH Terms: interventions — Phenylephrine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- phenylephrine (Experimental): 100 mcg of phenylephrine is administered at the time of reperfusion
  Interventions: Drug: phenylephrine
- epinephrine (Experimental): 10 mcg of epinephrine is administered iv at the time of reperfusion
  Interventions: Drug: epinephrine
- control (Placebo Comparator): 10 ml of normal saline is administered at the time of reperfusion
  Interventions: Drug: placebo control

INTERVENTIONS:
Drug: phenylephrine — 100 mcg of phenylephrine (volume 10 ml) iv at the time of reperfusion
  Arms: phenylephrine
Drug: epinephrine — 10mcg of epinephrine (volume 10 ml) is administered iv at the time of reperfusion
  Arms: epinephrine
Drug: placebo control — 10ml of normal saline is administered at the time of reperfusion
  Arms: control

SUMMARY:
Postreperfusion syndrome (PRS) is a relatively common phenomenon in patients undergoing liver transplantation which is characterized by an acute drop in blood pressure immediately after the prefusion is restored to the transplanted liver. We hypothesized that PRS would be prevented when phenylephrine or epinephrine is administered immediately prior to reperfusion in liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

- adults scheduled to undergo liver transplantation

Exclusion Criteria:

- pediatric liver transplantation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Ryu HG, Jung CW, Lee HC, Cho YJ. Epinephrine and phenylephrine pretreatments for preventing postreperfusion syndrome during adult liver transplantation. Liver Transpl. 2012 Dec;18(12):1430-9. doi: 10.1002/lt.23511. PMID 22821620

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 128 eligible candidates, 96 patients were enrolled in this study from Mar 2010 to Oct 2010 at SNUH.
Pre-assignment Details: Excluded(n=32) Children n=13 Coronary artery disease n=2 Valvular heart disease n=2 Atrial fibrillation n=1 Enrolled in other trial n=2 refusal to participate n=12
  Randomized (n=96) intraop portal vein rupture n=1 data recording error n=1 procedure failure n=1
  Analyzed n=93 (n=31 er each group)
Period: Overall Study
Arm/Group | Phenylephrine | Epinephrine | Control
Started | 31 | 33 | 32
Completed | 31 | 31 | 31
Not Completed | 0 | 2 | 1
Not completed — Physician Decision | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phenylephrine | Epinephrine | Control | Total
Number analyzed (Participants) | 31 | 33 | 32 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 27 | 31 | 29 | 87
  >=65 years | 4 | 2 | 3 | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (9) | 55 (10) | 52 (11) | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 7 | 26
  Male | 21 | 24 | 25 | 70
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 31 | 33 | 32 | 96

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Postreperfusion Syndrome (PRS)
Description: the number of patients who showed PRS (hypotension defined as < 30% of baseline mean arterial pressure [MAP] lasting over 1 min immediately after reperfusion of liver graft) was divided by the total number of patients enrolled for each group
Time Frame: immediately after reperfusion
Population: Initial assessment for eligibility: n=128 32 patients who did not meet the criteria were excluded 96 patients were randomized Contorol (32 patients) --> 1 patient was excluded because of portalvein rupture Epinephrine (33 patients) --> data recording error (1 patient) practice error (1 patient) Phenylephrine group (31 patient)
Measure: Number; unit: percentage of participants
Arm/Group | Phenylephrine | Epinephrine | Control
Number analyzed (Participants) | 31 | 31 | 31
percentage of participants | 45 | 39 | 87

ADVERSE EVENTS:
Arm/Group | Phenylephrine | Epinephrine | Control
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/31 | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No